CLINICAL TRIAL: NCT02889029
Title: Management of Complex Airway Stenoses With Dedicated Tailored Stents Wrought by 3D Computer-assisted Conception
Acronym: DASCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC31/15/7860
Record Dates: First submitted 2016-07-19; First posted 2016-09-05 (Estimated); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Obstructive Airway Disease
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- new 3D device (Experimental): dedicated tailored stents wrought by 3D computer-assisted conception
  Interventions: Device: new 3D device

INTERVENTIONS:
Device: new 3D device — dedicated tailored stents wrought by 3D computer-assisted conception

SUMMARY:
Management of complex airway stenoses with dedicated tailored stents wrought by 3D computer-assisted conception

Dedicated Airway Stents for Central Airway Stenoses

DASCAS

Toulouse University Hospital is the sponsor of this research.

This research will be conducted with the support of AnatomikModeling and ADERSPOT

* Background: Tracheobronchial stent are devices designed to manage central airway stenoses of various origins. Their shape and sizes are however not suitable for stenosis of complex anatomy.
* Purpose: The investigators propose to test the feasibility and safety of treating complex airway stenoses with dedicated tailored stents wrought by 3D computer-assisted conception

Abstract: Central airway obstruction is currently managed with non-personalized stents, which are usually efficient but lead to severe and potentially lethal complications in 10% of cases (stent migration, obstructive granuloma, perforation, hemoptysis). These stents seem particularly unsuited for anatomically complex stenosis.

Dedicated airway stents (wrought and tailored by 3D computer-assisted conception based on 3D chest CT-scan), by fitting perfectly tracheal or bronchial anatomy, should dramatically improve the tolerance and safety of such prostheses.

This first feasibility study, dedicated to patients suffering from anatomically complex stenosis will test the safety of treating patients with these new approach. It should lead to larger studies evaluating these new types of stents in larger indications.

After 3D computer-assisted modelization of airways, a virtual prosthesis and its shape are designed and the shape of the stent is wrought by 3D-machining by AnatomikModeling®. The stent is then build and sterilized by Sebbin® and inserted during rigid bronchoscopy on the same terms as pre-existing models.

Close follow up is then conducted, including clinical evaluation after one week, three and six months; spirometry at one week and 6 months and chest CT-scan at one week.

DETAILED DESCRIPTION:
Study design: Prospective monocentric feasibility study

Arm number or label and arm type: Only one experimental arm

Interventions:

After signature of a informed consent

Collection of clinical data (age, sex, etiology, site and mechanism of the stenosis, previous treatments dyspnea, quality of life (VQ11 questionnaire))

Chest CT-scan without contrast under continuous positive pressure

Spirometry (peak flow, FEV1)

Computer-assisted modelization of the shape of the prosthesis using 3D reconstruction of CT-scan

Machining of the shape in Ertacetal® (AnatomikModeling®)

Fabrication and sterilization of the stent in silicon (Sebbin®)

Insertion of the stent under rigid bronchoscopy and general anesthesia

Clinical follow-up at one week, 3 months and 6 months

Chest CT-scan without contrast at 1 week, spirometry at 1 week and 6 months

Number of subjects : 10 patients

Statistical analysis:

For the primary outcome, percentages of procedures conducted without complication at 1 week, 3 months, and 6 months and their confidence interval at 95% and incidences at 1 week, 3 months and 6 months for each complication will be calculated.

For secondary outcomes:

* Percentages of procedures conducted with improvement of dyspnea (improvement of at least one point of NYHA score) at 1 week, 3 months, and 6 months and their confidence interval at 95% will be calculated.
* Percentages of procedures conducted with improvement of quality of life (improvement of at least 10% of VQ11 score) at 1 week, 3 months, and 6 months and their confidence interval at 95% will be calculated.
* Percentages of procedures conducted with improvement of functional parameters (improvement of at least 20% of DEP or FEV1) at 1 week and 6 months and their confidence interval at 95% will be calculated.
* Percentage of procedures conducted with radiologic congruence of the stent at 1 week and its confidence interval at 95% will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Signature of the informed consent form
* Patient with a complex upper airway stenosis .
* Symptomatic stenosis ( Dyspnea > NYHA II , cough, PEF < 50%)
* Stenosis whose complex anatomy does not allow the establishment of a currently available stent on the market: the assessment of the experts ( consensus decision between 3 bronchoscopistes of interventional endoscopy service) or after failure of one or several models.
* Affiliated with a social security scheme

Exclusion Criteria:

* Indication of implementation of emergency aid : signs of acute respiratory distress , PEF < 20 % predicted , SpO2 oxygen saturation <90 % on room air
* Contraindication to rigid bronchoscopy (severe coagulation disorders not correct )
* Patient under legal protection system
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2020-11 (Actual)

PRIMARY OUTCOMES:
Change of percentage of procedures conducted without complications at 1 week , 3 months and 6 months | Change of percentage of procedures conducted without complications at 1 week, 3 months and 6 months
  percentages of procedures conducted without complication at 1 week, 3 months and 6 month and their confidence interval at 95% and incidences at 1 week, 3 months and 6 months for each complication will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Guibert, Dr, Principal Investigator — University Hospital, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guibert N, Didier A, Moreno B, Lepage B, Leyx P, Plat G, Mhanna L, Murris M, Mazieres J, Hermant C. Treatment of complex airway stenoses using patient-specific 3D-engineered stents: a proof-of-concept study. Thorax. 2019 Aug;74(8):810-813. doi: 10.1136/thoraxjnl-2018-212732. Epub 2019 Apr 3. PMID 30944151